CLINICAL TRIAL: NCT05347238
Title: Dopamine vs. Norepinephrine for Hypotension in Very Preterm Infants With Late-onset Sepsis: An International Comparative Effectiveness Research Project
Brief Title: Dopamine vs. Norepinephrine for Hypotension in Very Preterm Infants With Late-onset Sepsis
Status: Recruiting | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); The Hospital for Sick Children (Other); London Health Sciences Centre (Other); Windsor Regional Hospital (Other); Foothills Medical Centre (Other); Health Sciences Centre, Winnipeg, Manitoba (Other); St. Boniface Hospital (Other); Jewish General Hospital (Other); St. Justine's Hospital (Other); IWK Health Centre (Other); University College Cork (Other); Coombe Women and Infants University Hospital (Other); Island Health, Victoria, BC (Other); Assaf-Harofeh Medical Center (Other Government); Dayton Children's Hospital (Other); Banner University Medical Center (Other); Methodist Healthcare (Other); Hospital Universitario La Paz (Other); McMaster Children's Hospital (Other); Children's Hospital of Eastern Ontario (Other); BC Women's Hospital & Health Centre (Other); Stony Brook University (Other); The Children's Hospital at Montefiore (Other); Golisano Children's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: CTO 4009
Record Dates: First submitted 2022-04-12; First posted 2022-04-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Late-Onset Neonatal Sepsis; Extreme Prematurity; Neonatal Hypotension
MeSH Terms: conditions — Neonatal Sepsis | interventions — Dopamine; Norepinephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dopamine Units: Units who have standardized their practice with the use of Dopamine as a first line agent.
  Interventions: Drug: Dopamine
- Norepinephrine Units: Units who have standardized their practice with the use of Norepinephrine as a first line agent.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Dopamine — Start at 5mics/kg/min, increase every 16-30 minutes by 5 mics/kg/min to a maximum dose of 15 mics/kg/min or adequate response.
  Groups: Dopamine Units
Drug: Norepinephrine — Start at 0.05 mics/kg/min, increase every 16-30 minutes by 0.05 mics/kg/min to maximum dose of 0.15/mics/kg/min or adequate response
  Groups: Norepinephrine Units

SUMMARY:
Fluid-unresponsive hypotension needing cardiotropic drug treatment is a serious complication in very preterm neonates with suspected late-onset sepsis (LOS; defined as culture positive or negative bloodstream infection or necrotizing enterocolitis occurring >48 hours of age). In Canada, ~250 very preterm neonates receive cardiotropic drugs for LOS related fluid-unresponsive hypotension every year; of these ~35-40% die. Unlike for adult patients, there is little evidence to inform practice. While several medications are used by clinicians, the most frequently used medications are Dopamine (DA) and Norepinephrine (NE). However, their relative impact on patient outcomes and safety is not known resulting in significant uncertainty and inter- and intra-unit variability in practice. Conducting large randomized trials in this subpopulation can be operationally challenging and expensive. Comparative effectiveness research (CER), is a feasible alternative which can generate high-quality real-world evidence using real-world data, by comparing the impact of different clinical practices.

Aim: To conduct an international CER study, using a pragmatic clinical trial design, in conjunction with the existing infrastructure of the Canadian Neonatal Network to identify the optimal management of hypotension in very preterm neonates with suspected LOS.

Objective: To compare the relative effectiveness and safety of pharmacologically equivalent dosages of DA versus NE for primary pharmacotherapy for fluid-unresponsive hypotension in preterm infants born ≤ 32 weeks gestational age with suspected LOS.

Hypothesis: Primary treatment with NE will be associated with a lower mortality

Methods: This CER project will compare management approach at the unit-level allowing inclusion of all eligible patients admitted during the study period. 16 centers in Canada, 2 centers in Ireland, 1 center in each of Israel, Spain and the UK, and 6 centers in the United States have agreed to standardize their practice. All eligible patients deemed circulatory insufficient will receive fluid therapy (minimum 10-20 cc/kg). If hypotension remains unresolved:

Dopamine Units: start at 5mics/kg/min, increase every 16-30 minutes by 5 mics/kg/min to a maximum dose of 15 mics/kg/min or adequate response

Norepinephrine Units: start at 0.05 mics/kg/min, increase every 16-30 minutes by 0.05 mics/kg/min to maximum dose of 0.15/mics/kg/min or adequate response

DETAILED DESCRIPTION:
In this study, we will use real world data (RWD; defined as data generated during routine clinical practice) collected by our national Canadian Neonatal Network (CNN), which will be further expanded for this project.

The CNN is a well-established patient registry that includes members from 31 hospitals and 17 universities across Canada. The Network maintains a standardized NICU database and provides a unique opportunity for researchers to participate in collaborative projects. We will use the framework of Hypotheses Evaluating Treatment Effectiveness (HETE) research a form of comparative effectiveness research (CER).

Patient registries are emerging as a new method for assessment of treatments under the framework of CER. We will evaluate treatment effectiveness of two routinely used primary therapies for hypotension management in very preterm neonates with suspected LOS after standardizing treatment strategies and with a priori hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* ≤32 weeks gestational age and > 48 hours of life
* Receiving primary vasopressor therapy with Dopamine or Norepinephrine in the context of suspected late-onset sepsis or necrotizing enterocolitis with systemic hypotension (defined as: culture positive or negative bloodstream infection)

Exclusion Criteria:

* Known chromosomal or genetic anomalies
* Receiving primary therapy with agents other than Dopamine or Norepinephrine

Ages: 21 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All preterm infants born ≤32 weeks gestational age and > 48 hours of life with suspected sepsis with systemic hypotension admitted to the participating sites and meeting the above eligibility criteria will be included in the study.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
All cause in-hospital mortality | From illness onset to discharge (home or to another hospital) - assessed up to a maximum of 36 weeks after date of birth
  Death before discharge

SECONDARY OUTCOMES:
Episode-related death | <14 days from illness onset
  Episode-related death (yes or no- binary variable)
Treatment failure rate | 90 minutes after initial vasopressor initiation (or sooner if secondary dose added or primary agent replaced as per clinical discretion)
  Need for further dose escalation or use of additional agents (treatment failure = hypotension unresolved after reaching max dose (15mics/kg/min in Dopamine units and 0.15 mics/kg/min in Norepinephrine units)
New diagnosis of severe neurological injury | From illness onset to discharge (home or to another hospital) - assessed up to a maximum of 36 weeks after date of birth
  Grade III or Grade IV intraventricular hemorrhage or periventricular leukomalacia (yes or no- binary variable)
Bronchopulmonary dysplasia | Assessed at 36 weeks PMA
  Need for oxygen or positive pressure respiratory support at 36 weeks postmenstrual age (PMA) (yes or no- binary variable)
Retinopathy of prematurity | From illness onset to discharge (home or to another hospital) - assessed up to a maximum of 36 weeks after date of birth
  Diagnosis of retinopathy of prematurity - assessed by clinical staff (yes or no - binary variable)
Length of hospital stay | From admission date to discharge date - assessed up to a maximum of 36 weeks after date of birth
  Length of entire neonatal intensive care unit stay from admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Amish Jain, MBBS, MRCPCH, PhD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (23):
- United States (3):
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Dayton Children's Hospital, Dayton, Ohio
  - Methodist Healthcare, San Antonio, Texas
- Canada (16):
  - Foothill's Medical Centre, Calgary, Alberta
  - BC Women's Hospital, Vancouver, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - St.Boniface Hospital, Winnipeg, Manitoba
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - CHU Sainte- Justine, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
- Ireland (2):
  - University Cork College, Cork
  - Coombe Women & Infants University Hospital, Dublin
- Shamir Medical Center, Be’er Ya‘aqov, Israel
- La Paz University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No